CLINICAL TRIAL: NCT03250923
Title: CelAgace™ OraRinse (CAOR) Pilot Clinical Study for Management of Candidiasis Associated With Grade 0-II Mucositis
Brief Title: CelAgace™ OraRinse Solution for Treatment of Candidiasis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CelaCare Technologies, Inc. (Industry)
Collaborators: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2017-0042
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-02

CONDITIONS: Candidiasis, Oral
Keywords: Oral Candidiasis, Thrush, Oral Moniliasis
MeSH Terms: conditions — Candidiasis, Oral | interventions — acemannan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- silver citrate complex and acemannan (Experimental): This is a single arm open pilot trial. All participants will receive study drug.
  Interventions: Drug: silver citrate complex and acemannan

INTERVENTIONS:
Drug: silver citrate complex and acemannan — Oral rinse solution with each dose containing 100μg silver citrate complex and 40mg acemannan
  Other Names: CelAgace™ OraRinse Solution

SUMMARY:
CelAgace™ OraRinse (silver citrate complex and acemannan) Solution is planned to be evaluated for safety and effectiveness as a potential treatment for candidiasis, a yeast infection, commonly known as thrush, which is associated with mouth sores.

DETAILED DESCRIPTION:
CelAgace™ contains two active ingredients, a silver citrate complex salt (0.01mg/ml) that has demonstrated laboratory effectiveness against yeast organisms and acemannan (4.0mg/ml), a purified extract isolated from the inner leaf gel of the Aloe vera plant that has been used as a key ingredient in other oral care products. Patients will swish and spit the product 4 times daily (after meals and at bedtime) for 14 days. Following an initial office visit, patients will be evaluated on days 7 and 14 to determine response to the product.

ELIGIBILITY:
Inclusion Criteria:

* Radiation induced oral mucositis with resulting candidiasis
* Chemotherapy induced oral mucositis with resulting candidiasis
* Oral mucositis due to being immunocompromised with resulting candidiasis
* Stomatitis due to other causes with resulting candidiasis
* Currently have mild to moderate mucositis

Exclusion Criteria:

Patient:

* under the age of 18
* pregnant or breastfeeding
* inability to use an oral rinse
* hypersensitivity to Aloe Vera and/or Silver
* whose candida rinse culture was performed greater than 10 days prior to study entry.
* has any sort of removable dental appliance
* with previous or current history of any cancer of the oral cavity
* who received therapy for candidiasis within the past 30 days
* who used antifungal medication in the last 30 days
* who has severe to life threatening oral muositis (Grade III-IV) oral mucositis
* with impaired renal or hepatic function
* receiving high dose chemotherapy and total body irradiation in preparation for Hemopoietic Stem Cell Transplant (HSCT) or Concomitant use of Kepivance® (palifermin or rhKGF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Clinical cure as demonstrated by change and reduction from baseline in typical candida lesions and a negative candida rinse culture | Days 1(Baseline), 3, 7 and 14
  Rinse culture will be taken on Days 1, 7 and 14 to quantify Candidal Colony Forming Units and observational assessment will be done at study entry, Day 1, Days 3, 7, 14 using the WHO grading scale for response evaluation.

SECONDARY OUTCOMES:
Reduction in Pain | Days 1, 3, 7, 14
  Patients will complete a pain quality assessment rating scale (PQAS) during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline M. Plemons, DDS, MS, Principal Investigator — Texas A&M University College of Dentistry
Locations (1):
- Texas A&M University College of Dentistry, Dallas, Texas, United States